CLINICAL TRIAL: NCT04350073
Title: Longitudinal Energy Expenditure and Metabolic Effects in Patients With COVID-19 (LEEP-COVID)
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00105221
Record Dates: First submitted 2020-04-14; First posted 2020-04-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: COVID-19
Keywords: Respiratory failure; metabolic phenotype; mitochondrial phenotype; cardiometabolic phenotype; sarcopenia; malnutrition; critical care; muscle mass; cardiac function; heart failure; energy expenditure; nutrition; intensive care; COVID-19; SARS-CoV-2
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency; Sarcopenia; Malnutrition; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- COVID-19 ICU Patients: COVID-10 patients with respiratory failure admitted to the ICU
  Interventions: Device: Q-NRG Metobolic Cart Device; Device: MuscleSound Ultrasound; Device: Multifrequency Bioimpedance Spectroscopy
- ICU Patients (Control): Non-COVID-19 respiratory failure patients requiring mechanical ventilation > 48 h receiving similar ICU standards of care at Duke
  Interventions: Device: Q-NRG Metobolic Cart Device; Device: MuscleSound Ultrasound; Device: Multifrequency Bioimpedance Spectroscopy

INTERVENTIONS:
Device: Q-NRG Metobolic Cart Device — COVID-19 ICU patients will be measured using the Q-NRG device for up to 30 mins. These measurements will take place every other day while the patients are in the ICU. Then they will occur a minimum of 3 times a week until discharge.
Device: MuscleSound Ultrasound — COVID-19 ICU patients will have muscle mass, muscle glycogen, and muscle quality measured at rectus femoris (leg), intercostal, and temporal muscle. These measurements will take place every other day while the patients are in the ICU. Then they will occur a minimum of 3 times a week until discharge.
  Other Names: Muscle Mass Ultrasound
Device: Multifrequency Bioimpedance Spectroscopy — COVID-19 ICU patients will have body composition and phase angle measured using Multifrequency Bioimpedance Spectroscopy. These measurements will take place every other day while the patients are in the ICU. Then they will occur a minimum of 3 times a week until discharge.
  Other Names: InBody S10 BIA

SUMMARY:
This current proposal evaluates the Longitudinal Energy Expenditure and Metabolic Effects in Patients with COVID-19 (LEEP-COVID) to understand, guide and optimize our metabolic and nutritional care of these high risk patients. As no data exist for the metabolic effects of COVID-19 patients, this data is urgently needed and essential to assist in the care of COVID-19 patients worldwide. We are uniquely positioned at Duke to perform this research, as we are the only US center with 2 of the FDA-approved devices in existence currently capable of collecting this vital data to guide the care of COVID-19 patients worldwide.

DETAILED DESCRIPTION:
Currently, no longitudinal data exist describing the metabolic and cardiac effects of SARS-CoV-2 (COVID-19) infection. This data is urgently needed to assist in care and promote recovery of COVID-19 patients worldwide, and elderly patients who are at higher risk due to increased age, pre-existing risk factors (frailty, sarcopenia, malnutrition), and co-morbid conditions. Further, new pathologies such as COVID-19-related cardiac dysfunction must be described and rapidly identified. Our innovative measurements will provide direct non-invasive assessments of the effect of COVID-19 infection on key measures including energy expenditure, substrate utilization, muscle mass, cardiac function, mitochondrial function, and body composition. In addition, we will be able to provide objective data on key recovery intervention requirements including energy/nutritional requirements, effects of nutrition and rehabilitation efforts on muscle mass and energy state, and recovery of cardiac, muscle function.

Study Questions: We propose to evaluate longitudinal metabolic and cardiac pathophysiology in patients with COVID-19 to understand, guide and optimize our metabolic clinical care during acute hospitalization. Further, this data will be essential in providing objective data to guide physical recovery interventions including nutrition delivery and physical therapy to ensure functional recovery of COVID-19 patients.

We hypothesize: 1) COVID-19 will lead to significant, EE/metabolic changes, systemic mitochondrial dysfunction, significant muscle wasting and loss of function throughout the course of illness and during recovery. We hypothesize metabolic needs will initially decrease in acute illness and subsequently increase as patients transition from the acute phase of COVID illness to recovery phases. This data will guide nutrition and metabolic/clinical care in all phases of COVID-19 care where, for example, over-and under-feeding may pose risk to patient outcome. We hypothesize loss of muscle mass and physical function occurring in COVID-19 will significantly affect nutritional/rehabilitative/recovery of function/QoL needs and requires addressing to personalize care to optimize clinical and functional recovery efforts in older COVID-19 patients.

We believe longitudinal detailed indirect calorimetry with the innovative new Q-NRG device, cardiac assessment, body composition, and muscle and ultrasound measures in COVID-19 patients will play a key role in understanding and treating COVID-19 infection by providing objective data on the metabolic, cardiac, volume/fluid status, and nutrition needs of COVID-19 patients to the bedside clinician. This will increase our understanding of the pathophysiology of COVID-19 and the ability of clinical teams to optimize care and patient outcomes. These urgently needed data will lead to key advances in the clinical care of COVID-19 patients worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill COVID-19 patients greater or equal to 18 years of age patients requiring mechanical ventilation for > 48 hours who are admitted to Duke Surgical/Trauma ICU, Medical ICU, Cardiothoracic ICU, and Neuro ICU from admission to hospital discharge
* Patients must be enrolled within 72 hours of ICU admission
* Control: non-COVID-19 respiratory failure patients requiring mechanical ventilation > 48 h receiving similar ICU standards of care at Duke

Exclusion Criteria:

* Age less than 18 years old
* Fraction of inhaled oxygen (FIO2) > 70%
* Positive end expiratory pressure (PEEP) > 10cmH2O
* Peak ventilatory pressure > 30cmH20
* Presence of air leaks from thoracic drain tube
* Changes in vasoactive agent dose (>20%, <1 hr before or during IC)
* Agitation or change in sedative/analgesic dose (>20%, <1 hr before and/or during IC)
* Change in body temperature (>0.5°C, <1 hr before and/or during IC)
* Expected duration of ICU stay < 24 hours
* Expected survival of the patient < 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill COVID-19 or non-COVID-19 patients greater or equal to 18 years of age patients requiring mechanical ventilation for > 48 hours who are admitted to Duke Surgical/Trauma ICU, Medical ICU, Cardiothoracic ICU, and Neuro ICU from admission to hospital discharge
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-08-22 (Actual)

PRIMARY OUTCOMES:
Metabolic and Nutritional Needs of COVID-19 Patients: Measured by Changes of Resting Energy expenditure(REE) over time, as measured by the indirect calorimetry Q-NRG device | Minimum of every other day while in ICU (up to 10 days). Once discharged from ICU minimum of 3x a week until discharge (up to 3 weeks)
  The amount of CO2 produced combined with O2 consumed is called the REE (kcal/day) and is measured by the gases exchanged at the mouth.
Metabolic and Nutritional Needs of COVID-19 Patients:Changes of the Respiratory Exchange Ratio (RER) as measured by the indirect calorimetry Q-NRG device | Minimum of every other day while in ICU (up to 10 days). Once discharged from ICU minimum of 3x a week until discharge (up to 3 weeks)
  RER (ratio of CO2 produced to O2 consumed is called the respiratory exchange ratio (RER) and is measured by the gases exchanged at the mouth
Cardiac Output and Cardiac Measures (non-invasive) in COVID-19 patients | Minimum of every other day while in ICU (up to 10 days). Once discharged from ICU minimum of 3x a week until discharge (up to 3 weeks)
  Non-invasive, accurate calculation of cardiac output and other cardiac function measurements via Fick equation using direct measurement of VO2 & VCO2. As COVID-19 is known to have significant risk of cardiac failure & cardiac death this may allow early detection of cardiac changes that otherwise may not be recognized in these patients who will not routinely have invasive cardiac monitoring (I.e. Swan-Ganz catheter)

SECONDARY OUTCOMES:
Muscle Mass and Quality Changes from COVID-19: Measured via Changes of Intramuscular Adipose Tissue (IMAT) Content From CT Scans of the Psoas at the Level of L3/Th3 | Up to 1 year
  Measures the change over time of (standard of care) CT-derived area of intramuscular muscle mass and adipose tissue in cm2
Muscle Mass, Quality, Glycogen Changes in COVID-19: Via Metabolic/Muscle Imaging Derived From Muscle-Specific Ultrasound of Leg/Intercostal/Head Muscles | Every 3 days (+/- 1 day) while in ICU and then every 5 days (+/- 2 days) for the remainder of hospital stay. Maximum frequency, if requested by the clinical team (for the purposes of clinical care) can be up to once a day, every day.)
  The change over time of Ultrasound-derived muscle mass, muscle glycogen, and area of intramuscular adipose tissue in % and intramuscular glycogen content (IMGC) from rectus femurs - vastus laterals - intercostalis - temporalis - styloglossys
Body Composition in COVID-19 Patients: Measured via Multifrequency Bioimpedance Spectroscopy | Minimum of every other day while in ICU (up to 10 days). Once discharged from ICU minimum of 3x a week until discharge (up to 3 weeks)
Phase Angle in COVID-19 Patients: Measured via Multifrequency | Minimum of every other day while in ICU (up to 10 days). Once discharged from ICU minimum of 3x a week until discharge (up to 3 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Paul E Wischmeyer, MD, EDIC, FASPEN, FCCM, Principal Investigator — Duke University
Locations (1):
- Duke University Medial Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No